CLINICAL TRIAL: NCT03991559
Title: A Phase I, Two-arm, Open-label, Single-center, Dose-escalation Study to Evaluate the Safety, Tolerability and Recommended Dose and Delivery Mode of the Pan-immunotherapy in Subjects With Unresectable/ Metastatic Solid Tumors or Lymphomas
Brief Title: A Safety Study of the Pan-immunotherapy in Patients With Unresectable/Metastatic Solid Tumors or Lymphomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-039
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumor; Lymphoma
Keywords: anti-PD-1 antibody; Manganese; unresectable; metastatic
MeSH Terms: conditions — Lymphoma; Neoplasm Metastasis | interventions — manganese chloride; spartalizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-Escalation, intranasally (Active Comparator): With a standard 3+3 dose escalation design, the enrollment will proceed until the maximum tolerated dose (MTD) has been defined or the highest dose level has been reached.
  Interventions: Drug: Manganese Chloride; Drug: Anti-PD-1 antibody; Combination Product: Systemic therapy
- Dose-Escalation, inhalation (Active Comparator): With a standard 3+3 dose escalation design, the enrollment will proceed until the MTD has been defined or the highest dose level has been reached.
  Interventions: Drug: Manganese Chloride; Drug: Anti-PD-1 antibody; Combination Product: Systemic therapy

INTERVENTIONS:
Drug: Manganese Chloride — Administered intranasally in Arm 1 (0.05, 0.1 or 0.2 mg/kg/d) and by inhalation in Arm 2 (0.1, 0.2 or 0.4mg/kg/d) once daily in a 3-week cycle
Drug: Anti-PD-1 antibody — Administered intravenously, at 2-4mg/kg on day 3 in a 3-week cycle
  Other Names: Anti-PD-1 monoclonal antibody; PD-1 inhibitor
Combination Product: Systemic therapy — Whether and which should be given depends on the treatment regimen before enrollment.

SUMMARY:
Identification of T cell inhibitory signals, including PD-1/PD-L1, has prompted the development of a new class of cancer immunotherapy that could restore an adequate immunosurveillance against the neoplasm and enhance T-cell-mediated anticancer immune responses. However, elimination of cancer by T cells is only one step in the Cancer-Immunity Cycle, which enable providing several therapeutic targets and tailoring of combinations of immune therapies. Manganese has been confirmed to activate antigen-presenting cells and function as mucosal immunoadjuvants in pre-clinical studies. This study is a first-in-man, Phase I, 3 + 3 dose escalation study of a combined regimen of Manganese and anti-PD-1 antibody with or without chemotherapies in subjects with unresectable/ metastatic solid tumors or lymphomas. This study is designed to assess the safety, tolerability, pharmacokinetic profile (PK profile), mode of delivery and Recommended Phase 2 Dose (RP2D) of this regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically proven unresectable/ metastatic solid tumors or lymphomas.
2. ≥ 18 years old.
3. Life expectancy of at least 6 months.
4. Eastern Cooperative Oncology Group performance status 0-2.
5. Subjects must have at least one measurable lesion ≥ 1 cm as defined by response criteria.
6. Subjects must have received at least two frontline therapies, except for patients initially diagnosed with local advanced or metastatic pancreatic cancer or cholangiocarcinoma.
7. Subjects must be off prior therapy for at least 4 weeks prior to Day 1. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months. Subjects with Anti-PD-1 antibody are eligible which must be resistance.
8. Adequate organ function.
9. Participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. T cell lymphomas or leukemia.
4. Prior organ allograft.
5. Women who are pregnant or breastfeeding.
6. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
7. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment-related adverse events (AEs) | Approximately 6 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0. AEs were considered to be treatment-related if they had started or worsened within the interval from first study drug administration until the follow-up visit.
Number of subjects with specific Manganese-related adverse events | Approximately 6 months
  Manganese-related AEs were considered to be that start or worsen after administration Manganese administration，improve after withdrawal, and even occur again after re-administration.

SECONDARY OUTCOMES:
Preliminary efficacy evaluation | Approximately 6 months
  Objective response rate (ORR) and disease control rate (DCR) will be evaluated by investigators per the RECIST V1.1.
The q3w pharmacokinetic profile of Manganese | Approximately 3 months
  PK parameters such as Maximum concentration (Cmax) are assessed.
Number of participants with laboratory test abnormalities | Approximately 3 months
  The laboratory tests of serum cytokines and chemokines will be performed on day 1 and 3 of each cycle, and the abnormality will be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China